CLINICAL TRIAL: NCT04822064
Title: Comparison of Oral Chloral Hydrate and Combination of Intranasal Dexmedetomidine and Ketamine for Rescue After Failed Pediatric Procedural Sedation: a Randomized Controlled Trial
Brief Title: Comparison of Oral Chloral Hydrate and Combination of Intranasal Dexmedetomidine and Ketamine for Rescue After Failed Pediatric Procedural Sedation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IN DEXKET rescue
Record Dates: First submitted 2021-03-19; First posted 2021-03-30 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Sedation
Keywords: pediatric; procedural sedation; chloral hydrate; intranasal dexmedetomidine; intranasal ketamine
MeSH Terms: interventions — Ketamine; Chloral Hydrate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intranasal dexmedetomdine and kemtaine (Experimental): Additional intranasal administration of dexmedetomidine (2mcg/kg) and ketamine (3mg/kg) to induce rescue sedation (pediatric sedation state scale = 1,2,3) after failed sedation attempt (PSSS=4,5) with oral chloral hydrate (50mg/kg)
  Interventions: Drug: Intranasal dexmedetomidine and ketamine
- oral chloral hydrate (Active Comparator): Additional oral chloral hydrate (50mg/kg) administration to induce rescue sedation (pediatric sedation state scale = 1,2,3) after failed sedation attempt (PSSS=4,5) with oral chloral hydrate (50mg/kg)
  Interventions: Drug: Oral chloral hydrate

INTERVENTIONS:
Drug: Intranasal dexmedetomidine and ketamine — Additional intranasal administration of dexmedetomidine (2mcg/kg) and ketamine (3mg/kg) to induce rescue sedation (pediatric sedation state scale = 1,2,3) after failed sedation attempt (PSSS=4,5) with oral chloral hydrate (50mg/kg)
  Arms: intranasal dexmedetomdine and kemtaine
Drug: Oral chloral hydrate — Additional oral chloral hydrate (50mg/kg) administration to induce rescue sedation (pediatric sedation state scale = 1,2,3) after failed sedation attempt (PSSS=4,5) with oral chloral hydrate (50mg/kg)
  Arms: oral chloral hydrate

SUMMARY:
In Korea, oral chloral hydrate is still widely used for pediatric procedural sedation. The primary objective of the study is to evaluate the effect of intranasal dexmedetomidine (2mcg/kg) and ketamine (3mg/kg) on the success rate of rescue sedation after failed sedation (PSSS=4,5) with chloral hydrate (50mg/kg) The hypothesis of this study is that the intranasal dexmedetomidine (2mcg/kg) and ketamine (3mg/kg) will improve the success rate of rescue sedation (PSSS=1,2,3) within 15 minutes. This is a prospective, parallel-arm, single-blinded, multi-center, randomized controlled trial comparing the effect of intranasal dexmedetomidine (2mcg/kg) and ketamine (3mg/kg) with oral chloral hydrate (50mg/kg) in pediatric patients after failed sedation attempt with oral chloral hydrate. Prior to the procedure, each patient will be randomized in the control arm (oral chloral hydrate) or study arm (intranasal dexmedetomidine and ketamine).

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients who need procedural sedation (Age < 7 years)
* ASA (American Society of Anesthesiologists) physical status 1-3
* Failed to induce sedation with oral chloral hydrate 50mg/kg

Exclusion Criteria:

* ASA (American Society of Anesthesiologists) physical status 4-5
* History of hypersensitivity to Dexmedetomidine, Ketamine, or Chloral hydrate
* Recent administration of Alpha 2 adrenergic receptor agonist or antagonist
* Cannot administrate oral medication (e.g. Swallowing difficulty)
* Cannot administrate intranasal medication(e.g. Excessive rhinorrhea)
* Unstable vital signs, Unstable arrhythmia

Max Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Success rate of adequate rescue sedation (PSSS = 1, 2, 3) within 15 minutes % | During pediatric procedural sedation (up to 1 hour)
  Success rate of adequate rescue sedation (Pediatric Sedation State Scale= 1,2,3) within 15 minutes after sedative administration. %

SECONDARY OUTCOMES:
Onset time of rescue sedation (PSSS =1,2,3) (min) | During pediatric procedural sedation (up to 3 hour)
  Onset time of rescue sedation (Pediatric Sedation State Scale= 1,2,3) after rescue sedative administration.
Duration of rescue sedation = Recovery time (PSSS =4,5) | During pediatric procedural sedation (up to 3 hour)
  Pediatric Sedation State Scale= 4,5 after recovery of sedation
PSSS(Pediatric Sedation State Scale, 0-5) | During pediatric procedural sedation (up to 3 hour)
  5 Patient is moving in a manner that impedes the proceduralist and requires forceful immobilization.
  4 Moving during the procedure that requires gentle immobilization for positioning.
  3 Expression of pain or anxiety on face, but not moving or impeding completion of the procedure.
  2 Quiet (asleep or awake), not moving during procedure, and no frown (or brow furrow) indicating pain or anxiety.
  1 Deeply asleep with normal vital signs, but requiring airway intervention and/or assistance 0 Sedation associated with abnormal physiologic parameters that require acute intervention q 10min
HR during sedation (/min) | During pediatric procedural sedation (up to 3 hour)
  HR(/min) at Baseline(T0), q 10min
SpO2 during sedation (%) | During pediatric procedural sedation (up to 3 hour)
  SpO2(%) by pulse oximetry at Baseline(T0), q 10min
Respiratory rate during sedation (/min) | During pediatric procedural sedation (up to 3 hour)
  RR(/min) at Baseline(T0), q 10min
the incidence of PSSS=0 (Abnormal physiologic parameter that require acute intervention) % | During pediatric procedural sedation (up to 3 hour)
  the incidence of PSSS=0 (Abnormal physiologic parameter that require acute intervention) %
The incidence of respiratory intervention: Manual ventilation or Artificial airway % | During pediatric procedural sedation (up to 3 hour)
  The incidence of respiratory intervention: Manual ventilation or Artificial airway %
The incidence of significant desaturation (SpO2 < 95% or -10% from baseline, >10 seconds) % | During pediatric procedural sedation (up to 3 hour)
  The incidence of significant desaturation (SpO2 < 95% or -10% from baseline, >10 seconds) %
The incidence of significant apnea (>20seconds) % | During pediatric procedural sedation (up to 3 hour)
  The incidence of significant apnea (>20seconds) %
The lowest SpO2 value (%) | During pediatric procedural sedation (up to 3 hour)
  The lowest SpO2 value (%)
The incidence of hemodynamic intervention: fluid management, intravenous medication % | During pediatric procedural sedation (up to 3 hour)
  The incidence of hemodynamic intervention: fluid management, intravenous medication %
The incidence of significant bradycardia (-30% from baseline) % | During pediatric procedural sedation (up to 3 hour)
  The incidence of significant bradycardia (-30% from baseline) %
The incidence of significant hypotension (-30% from baseline) % | During pediatric procedural sedation (up to 3 hour)
  The incidence of significant hypotension (-30% from baseline) %
Patients' acceptance (1=excellent, 2=good, 3=fair, 4=poor) | During pediatric procedural sedation (up to 3 hour)
  Patients' acceptance (1=excellent, 2=good, 3=fair, 4=poor)
Separation anxiety (1=easy, 2=whimper, 3=cry, 4=cry and cling to parents) | During pediatric procedural sedation (up to 3 hour)
  Separation anxiety (1=easy, 2=whimper, 3=cry, 4=cry and cling to parents)
Physicians' satisfaction (1=excellent, 2=good, 3=fair, 4=poor) | During pediatric procedural sedation (up to 3 hour)
  Physicians' satisfaction (1=excellent, 2=good, 3=fair, 4=poor)
The incidence of Other side effects (Ex: Nausea/Vomit, Allergic reaction, Etc) | During pediatric procedural sedation (up to 3 hour)
  The incidence of Other side effects (Ex: Nausea/Vomit, Allergic reaction, Etc)
The incidence of Rescue sedation failure (PSSS =0,4,5) after 30 min % | During pediatric procedural sedation (up to 3 hour)
  The incidence of Rescue sedation failure (PSSS =0,4,5) after 30 min %
The incidence of Completion of procedure | During pediatric procedural sedation (up to 3 hour)
  The incidence of Completion of procedure
Total cost of sedation (KRW) | During pediatric procedural sedation (up to 1 day)
  Total cost of sedation (KRW)

CONTACTS AND LOCATIONS:
Locations (1):
- Jin-Tae Kim, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang W, Wang Z, Song X, Fan Y, Tian H, Li B. Comparison of rescue techniques for failed chloral hydrate sedation for magnetic resonance imaging scans--additional chloral hydrate vs intranasal dexmedetomidine. Paediatr Anaesth. 2016 Mar;26(3):273-9. doi: 10.1111/pan.12824. Epub 2015 Dec 30. PMID 26714442
- [Background] Cao Q, Lin Y, Xie Z, Shen W, Chen Y, Gan X, Liu Y. Comparison of sedation by intranasal dexmedetomidine and oral chloral hydrate for pediatric ophthalmic examination. Paediatr Anaesth. 2017 Jun;27(6):629-636. doi: 10.1111/pan.13148. Epub 2017 Apr 17. PMID 28414899
- [Background] Sheta SA, Al-Sarheed MA, Abdelhalim AA. Intranasal dexmedetomidine vs midazolam for premedication in children undergoing complete dental rehabilitation: a double-blinded randomized controlled trial. Paediatr Anaesth. 2014 Feb;24(2):181-9. doi: 10.1111/pan.12287. Epub 2013 Nov 15. PMID 24237879
- [Background] Zanaty OM, El Metainy SA. A comparative evaluation of nebulized dexmedetomidine, nebulized ketamine, and their combination as premedication for outpatient pediatric dental surgery. Anesth Analg. 2015 Jul;121(1):167-171. doi: 10.1213/ANE.0000000000000728. PMID 25822924
- [Background] Zhang W, Fan Y, Zhao T, Chen J, Zhang G, Song X. Median Effective Dose of Intranasal Dexmedetomidine for Rescue Sedation in Pediatric Patients Undergoing Magnetic Resonance Imaging. Anesthesiology. 2016 Dec;125(6):1130-1135. doi: 10.1097/ALN.0000000000001353. PMID 27627818
- [Background] Jun JH, Kim KN, Kim JY, Song SM. The effects of intranasal dexmedetomidine premedication in children: a systematic review and meta-analysis. Can J Anaesth. 2017 Sep;64(9):947-961. doi: 10.1007/s12630-017-0917-x. Epub 2017 Jun 21. PMID 28639236
- [Background] Abdel-Ghaffar HS, Kamal SM, El Sherif FA, Mohamed SA. Comparison of nebulised dexmedetomidine, ketamine, or midazolam for premedication in preschool children undergoing bone marrow biopsy. Br J Anaesth. 2018 Aug;121(2):445-452. doi: 10.1016/j.bja.2018.03.039. Epub 2018 Jun 22. PMID 30032884
- [Background] Poonai N, Canton K, Ali S, Hendrikx S, Shah A, Miller M, Joubert G, Rieder M, Hartling L. Intranasal ketamine for procedural sedation and analgesia in children: A systematic review. PLoS One. 2017 Mar 20;12(3):e0173253. doi: 10.1371/journal.pone.0173253. eCollection 2017. PMID 28319161